CLINICAL TRIAL: NCT03185130
Title: Intravenous Fluids in Benign Headaches Trial: A Randomized Single Blind Clinical Trial
Brief Title: Intravenous Fluids in Benign Headaches Trial
Acronym: I-FiBH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center of Southern Nevada (Other)
Responsible Party: Principal Investigator, Joseph (Tony) Zitek, MD, MD, University Medical Center of Southern Nevada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-54
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Headache
Keywords: Headache; Benign Headache
MeSH Terms: conditions — Headache | interventions — Saline Solution; Sodium Chloride; Prochlorperazine; Diphenhydramine

STUDY DESIGN:
Intervention Model Description: This will be a single center, prospective, single blinded randomized controlled trial on a convenience sample of patients presenting to the adult or pediatric ED with a chief complaint of headache.
Who Masked: Participant
Masking Description: By necessity the subject will be blinded but the RN administering the IV fluids will need to know the rate of infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Treatment Arm (Active Comparator): Standard Treatment Arm will receive: normal saline at 5 ml IV given over 1 hour, prochlorperazine 0.15 mg/kg up to 10 mg IV, diphenhydramine 1mg/kg (up to 50 mg) IV.
  Interventions: Drug: Normal Saline 5mL; Drug: Prochlorperazine 0.15 mg/kg up to 10 mg IV; Drug: Diphenhydramine 1 mg/kg up to 50 mg IV
- Study Arm (Experimental): Study arm patients will receive: normal saline at 20 mL/kg (up to 1000 mL) given over 1 hour, prochlorperazine 0.15 mg/kg up to 10 mg IV, diphenhydramine 1mg/kg (up to 50 mg) IV.
  Interventions: Drug: Normal Saline 20mL/kg; Drug: Prochlorperazine 0.15 mg/kg up to 10 mg IV; Drug: Diphenhydramine 1 mg/kg up to 50 mg IV

INTERVENTIONS:
Drug: Normal Saline 5mL — Control arm subjects will receive Normal Saline 5 mL IV over 1 hour
  Other Names: NS; Saline
  Arms: Standard Treatment Arm
Drug: Normal Saline 20mL/kg — Study arm subjects will receive Normal Saline 20 mL/kg IV (up to 1000 mL) given IV over 1 hour,
  Other Names: NS; Saline
  Arms: Study Arm
Drug: Prochlorperazine 0.15 mg/kg up to 10 mg IV — Standard Treatment Arm and Study Arm will receive prochlorperazine 0.15 mg/kg up to 10mg IV slow push
  Other Names: Compazine
Drug: Diphenhydramine 1 mg/kg up to 50 mg IV — Diphenhydramine dose 1 mg/kg up to 50 mg IV slow push
  Other Names: Benadryl

SUMMARY:
Migraine headache has a 1-year period prevalence in the US of 11.7% and accounts for approximately 1.2 million migraine visits to US emergency departments per year . There are numerous studies that discuss treatment for migraine and other benign headaches within the emergency department (ED), however, there are very few that discuss specifically the use of intravenous fluids (IVF) for headache treatment. Many of these studies look at various options for treating migraine and other benign headaches: treatment options include dopamine antagonists, opioids, non-steroid anti-inflammatory drugs (NSAIDs), triptans, anti-epileptics and ergot derivatives. Comparisons have been done between many of these treatment options with dopamine antagonists appearing to be the most effective, compared to other treatments The dopamine antagonist with the most evidence and availability for benign headaches is prochlorperazine. Given that IVF administration is a common part of treatment regimen for benign headache patients in the emergency department and given the lack of randomized trials in adults, the investigators aim to study the use of IVF on pain reduction in headache patients in the adult ED. There has been one randomized trial in pediatrics that shows IVF may help in patients with migraines, whereas the adult literature has no randomized control trials and a review of data shows that fluids do not help relieve pain in migraine headache patients. This study will include both adult and pediatric patients presenting to the Emergency Department with complaint of benign headache.

DETAILED DESCRIPTION:
This will be a single center, prospective, single blinded randomized controlled trial on a convenience sample of patients presenting to the adult or pediatric ED with a chief complaint of headache. Subjects will only be enrolled when a physician or research assistant who is familiar with the study protocol is available to enroll patients. Written, informed consent will be obtained from each patient. Consent will include a discussion of the risks and benefits. In addition to parental informed consent in the pediatric population, age appropriate verbal assent will be obtained from pediatric subjects. After 30 minutes, the treating provider will be permitted to administer a "rescue medication" of their choice for further treatment. If there is an untoward event that requires the patient to know which IVF dose was administered, patient will unblinded and will not continue in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10 to 65 years
2. Temperature less than 100.4 F
3. Normal neurologic exam and normal mental status

Exclusion Criteria:

1. Pregnant
2. Meningeal signs are present
3. Acute angle closure glaucoma is suspected
4. Head trauma within the previous two weeks
5. Lumbar puncture within the previous two weeks
6. Thunderclap onset of the headache
7. Known allergy to one of the study drugs
8. History of intracranial hypertension
9. Is a prisoner
10. Patient declined informed consent
11. Non-English speaking patient or parent/guardian for pediatric patients
12. Attending provider excludes patient
13. Severe Dehydration

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Zitek, MD, Principal Investigator — University Medical Center of Southern Nevada
Locations (1):
- University medical Center of Southern Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared.

REFERENCES:
- [Background] Lipton RB, Bigal ME, Diamond M, Freitag F, Reed ML, Stewart WF; AMPP Advisory Group. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology. 2007 Jan 30;68(5):343-9. doi: 10.1212/01.wnl.0000252808.97649.21. PMID 17261680
- [Background] Friedman BW, West J, Vinson DR, Minen MT, Restivo A, Gallagher EJ. Current management of migraine in US emergency departments: an analysis of the National Hospital Ambulatory Medical Care Survey. Cephalalgia. 2015 Apr;35(4):301-9. doi: 10.1177/0333102414539055. Epub 2014 Jun 19. PMID 24948146
- [Background] Balbin JE, Nerenberg R, Baratloo A, Friedman BW. Intravenous fluids for migraine: a post hoc analysis of clinical trial data. Am J Emerg Med. 2016 Apr;34(4):713-6. doi: 10.1016/j.ajem.2015.12.080. Epub 2015 Dec 30. PMID 26825817
- [Background] Cicek M, Karcioglu O, Parlak I, Ozturk V, Duman O, Serinken M, Guryay M. Prospective, randomised, double blind, controlled comparison of metoclopramide and pethidine in the emergency treatment of acute primary vascular and tension type headache episodes. Emerg Med J. 2004 May;21(3):323-6. doi: 10.1136/emj.2002.000356. PMID 15107371
- [Background] Friedman BW, Adewunmi V, Campbell C, Solorzano C, Esses D, Bijur PE, Gallagher EJ. A randomized trial of intravenous ketorolac versus intravenous metoclopramide plus diphenhydramine for tension-type and all nonmigraine, noncluster recurrent headaches. Ann Emerg Med. 2013 Oct;62(4):311-318.e4. doi: 10.1016/j.annemergmed.2013.03.017. Epub 2013 Apr 6. PMID 23567060
- [Background] Kostic MA, Gutierrez FJ, Rieg TS, Moore TS, Gendron RT. A prospective, randomized trial of intravenous prochlorperazine versus subcutaneous sumatriptan in acute migraine therapy in the emergency department. Ann Emerg Med. 2010 Jul;56(1):1-6. doi: 10.1016/j.annemergmed.2009.11.020. Epub 2010 Jan 4. PMID 20045576
- [Background] Tanen DA, Miller S, French T, Riffenburgh RH. Intravenous sodium valproate versus prochlorperazine for the emergency department treatment of acute migraine headaches: a prospective, randomized, double-blind trial. Ann Emerg Med. 2003 Jun;41(6):847-53. doi: 10.1067/mem.2003.195. PMID 12764341
- [Background] Jones J, Sklar D, Dougherty J, White W. Randomized double-blind trial of intravenous prochlorperazine for the treatment of acute headache. JAMA. 1989 Feb 24;261(8):1174-6. PMID 2915441
- [Background] Friedman BW, Esses D, Solorzano C, Dua N, Greenwald P, Radulescu R, Chang E, Hochberg M, Campbell C, Aghera A, Valentin T, Paternoster J, Bijur P, Lipton RB, Gallagher EJ. A randomized controlled trial of prochlorperazine versus metoclopramide for treatment of acute migraine. Ann Emerg Med. 2008 Oct;52(4):399-406. doi: 10.1016/j.annemergmed.2007.09.027. Epub 2007 Nov 19. PMID 18006188
- [Background] Callan JE, Kostic MA, Bachrach EA, Rieg TS. Prochlorperazine vs. promethazine for headache treatment in the emergency department: a randomized controlled trial. J Emerg Med. 2008 Oct;35(3):247-53. doi: 10.1016/j.jemermed.2007.09.047. Epub 2008 Jun 5. PMID 18534808
- [Background] Coppola M, Yealy DM, Leibold RA. Randomized, placebo-controlled evaluation of prochlorperazine versus metoclopramide for emergency department treatment of migraine headache. Ann Emerg Med. 1995 Nov;26(5):541-6. doi: 10.1016/s0196-0644(95)70001-3. PMID 7486359
- [Background] Miner JR, Fish SJ, Smith SW, Biros MH. Droperidol vs. prochlorperazine for benign headaches in the emergency department. Acad Emerg Med. 2001 Sep;8(9):873-9. doi: 10.1111/j.1553-2712.2001.tb01147.x. PMID 11535479
- [Background] Dychter SS, Gold DA, Carson D, Haller M. Intravenous therapy: a review of complications and economic considerations of peripheral access. J Infus Nurs. 2012 Mar-Apr;35(2):84-91. doi: 10.1097/NAN.0b013e31824237ce. PMID 22382792
- [Background] Homer LD, Holmes KR. Risks associated with 72- and 96-hour peripheral intravenous catheter dwell times. J Intraven Nurs. 1998 Sep-Oct;21(5):301-5. PMID 9814284
- [Background] Gentges J, Arthur A, Stamile T, Figureido M. Peripheral Intravenous Line Placement and Utilization in an Academic Emergency Department. J Emerg Med. 2016 Feb;50(2):235-8. doi: 10.1016/j.jemermed.2015.08.006. PMID 26433429
- [Background] Myburgh JA. Fluid resuscitation in acute medicine: what is the current situation? J Intern Med. 2015 Jan;277(1):58-68. doi: 10.1111/joim.12326. Epub 2014 Nov 25. PMID 25352314
- [Background] Tfelt-Hansen P, Pascual J, Ramadan N, Dahlof C, D'Amico D, Diener HC, Hansen JM, Lanteri-Minet M, Loder E, McCrory D, Plancade S, Schwedt T; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: third edition. A guide for investigators. Cephalalgia. 2012 Jan;32(1):6-38. doi: 10.1177/0333102411417901. No abstract available. PMID 22384463
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299
- [Background] Patniyot IR, Gelfand AA. Acute Treatment Therapies for Pediatric Migraine: A Qualitative Systematic Review. Headache. 2016 Jan;56(1):49-70. doi: 10.1111/head.12746. PMID 26790849
- [Background] Richer L, Craig W, Rowe B. Randomized controlled trial of treatment expectation and intravenous fluid in pediatric migraine. Headache. 2014 Oct;54(9):1496-505. doi: 10.1111/head.12443. Epub 2014 Aug 28. PMID 25168404
- [Derived] Zitek T, Sigal T, Sun G, Martin Manuel C, Tran K. I-FiBH trial: intravenous fluids in benign headaches-a randomised, single-blinded clinical trial. Emerg Med J. 2020 Aug;37(8):469-473. doi: 10.1136/emermed-2019-209389. Epub 2020 Jul 3. PMID 32620543

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Treatment Arm | Study Arm
Started | 23 | 35
Completed | 23 | 33
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment Arm | Study Arm | Total
Number analyzed (Participants) | 23 | 35 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (14.7) | 32.3 (14.1) | 32.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 6 | 15 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 12 | 17
  Not Hispanic or Latino | 18 | 23 | 41
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 35 | 58

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Pain Scores at 60 Minutes
Description: The primary outcome measure will be the mean reduction in pain scores at 60 min. In other words the pain score at time zero minus the pain score at time 60 minutes. Pain scores are measured 0-100, with 0 being no pain and 100 being maximal pain, on a visual analog scale score. Higher numbers indicate more pain reduction.
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: reduction in visual analog pain score
Arm/Group | Standard Treatment Arm | Study Arm
Number analyzed (Participants) | 23 | 33
reduction in visual analog pain score | 48.7 (29.3) | 48.3 (31.0)

2. Secondary Outcome: Reduction in Pain Score at 30 Minutes
Description: The mean reduction in pain scores at 30 minutes. This is calculated as the pain score at time zero minus the pain score at time 30 minutes. Pain scores are measured 0-100 on a visual analog scale score, with 0 being no pain and 100 being maximal pain. Higher numbers indicate more pain reduction.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: change in pain score
Arm/Group | Standard Treatment Arm | Study Arm
Number analyzed (Participants) | 23 | 35
change in pain score | 34.8 (29.6) | 31.8 (27.1)

3. Secondary Outcome: Admissions
Description: The difference between the rates of admission will be measured.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Arm | Study Arm
Number analyzed (Participants) | 23 | 35
Participants | 0 | 2

4. Secondary Outcome: Reduction in Nausea Score at 60 Minutes
Description: The reduction in mean nausea scores will be measured. This is calculated as the nausea score at time zero minus the nausea score at time 60 minutes. Nausea is measured from 0-100 on a visual analog scale with 0 being no nausea and 100 being maximal nausea. Higher numbers indicate more reduction in nausea.
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: reduction in nausea score
Arm/Group | Standard Treatment Arm | Study Arm
Number analyzed (Participants) | 23 | 33
reduction in nausea score | 31.8 (33.4) | 25.2 (34.2)

5. Secondary Outcome: Vomiting
Description: The difference in the percentage of patients in each group who vomit within one hour after the treatment starts.
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Arm | Study Arm
Number analyzed (Participants) | 23 | 33
Participants | 0 | 0

6. Secondary Outcome: Rescue Medication
Description: The difference between the percentage of patients requiring rescue medications for headache will be measured. "Rescue medications" are defined as any medication administered to the patient in the emergency department for their headache after the initial medications.
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Arm | Study Arm
Number analyzed (Participants) | 23 | 35
Participants | 3 | 7

7. Secondary Outcome: Percentage of Patients With Persistent Headache
Description: The difference between the rates of persistent headache with telephone follow up.
Time Frame: 24-48 hours after discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Arm | Study Arm
Number analyzed (Participants) | 17 | 27
Participants | 4 | 11

ADVERSE EVENTS:
Time Frame: 48 hours
Groups:
- Standard Treatment Arm: Standard Treatment Arm will receive: normal saline at 5 ml IV given over 1 hour, prochlorperazine 0.15 mg/kg up to 10 mg IV, diphenhydramine 1mg/kg (up to 50 mg) IV.
  Normal Saline 5mL: Control arm subjects will receive Normal Saline 5 mL IV over 1 hour
  Prochlorperazine 0.15 mg/kg up to 10 mg IV: Standard Treatment Arm and Study Arm will recieve prochlorperazine 0.15 mg/kg up to 10mg IV slow push
  Diphenhydramine 1 mg/kg up to 50 mg IV: Diphenhydramine dose 1 mg/kg up to 50 mg IV slow push
- Study Arm: Study arm patients will receive: normal saline at 20 mL/kg (up to 1000 mL) given over 1 hour, prochlorperazine 0.15 mg/kg up to 10 mg IV, diphenhydramine 1mg/kg (up to 50 mg) IV.
  Normal Saline 20mL/kg: Study arm subjects will receive Normal Saline 20 mL/kg IV (up to 1000 mL) given IV over 1 hour,
  Prochlorperazine 0.15 mg/kg up to 10 mg IV: Standard Treatment Arm and Study Arm will recieve prochlorperazine 0.15 mg/kg up to 10mg IV slow push
  Diphenhydramine 1 mg/kg up to 50 mg IV: Diphenhydramine dose 1 mg/kg up to 50 mg IV slow push
Arm/Group | Standard Treatment Arm | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/35
Other Adverse Events (participants affected / at risk) | 0/23 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03185130/Prot_SAP_000.pdf